CLINICAL TRIAL: NCT04351971
Title: Immediate Effects of the C0-C1 Mobilization Technique on Upper Cervical Mobility and Pressure Threshold in Patients With Chronic Neck Pain
Brief Title: Immediate Effects of the C0-C1 Mobilization Technique in Patients With Chronic Neck Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad San Sebastián (Other)
Responsible Party: Principal Investigator, gonzalo arias alvarez, Principal Investigator, Universidad San Sebastián
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1909-91
Record Dates: First submitted 2020-04-10; First posted 2020-04-17 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Musculoskeletal Manipulations; Cervical Pain
Keywords: manual therapies; Chronic Pain; Range of Motion
MeSH Terms: conditions — Neck Pain; Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Study participants will be assigned a random number and will be divided into two research groups (control group and intervention group). In this sense, both the patient and the therapist in charge of carrying out the evaluation will not know which group each subject belongs to.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The dorsal sliding technique C0-C1 will be applied to this group.
  Interventions: Other: Intervention Group
- Placebo group (Sham Comparator): A placebo dorsal mobilization technique will be applied
  Interventions: Other: Placebo group

INTERVENTIONS:
Other: Intervention Group — The patient's position is in the supine position. The therapist identifies the arches of the atlas and positions one hand at this level with the fingers extended. The other hand is located in the occipital region. Subsequently, the therapist makes a pressure with his shoulder assessing the movement and applies a pressure to the back. This technique is performed by mobilization cycles of 15 seconds and 3 seconds of rest for a total period of 5 minutes.The patient's position is in the supine position. The therapist identifies the arches of the atlas and positions one hand at this level with the fingers extended. The other hand is located in the occipital region. Subsequently, the therapist makes a pressure with his shoulder assessing the movement and applies a pressure to the back. This technique is performed by mobilization cycles of 15 seconds and 3 seconds of rest for a total period of 5 minutes.
  Arms: Intervention Group
Other: Placebo group — The technique consists of placing the patient in the supine position, one hand is located in the arches of the atlas, the other hand is located in the occipital. The therapist's shoulder is located in the anterior region. This position is maintained for 5 minutes without exerting pressure.
  Arms: Placebo group

SUMMARY:
Background: Skeletal muscle-type pain is one of the main reasons for consultations in health centers. In Chile, it is estimated that the prevalence reaches 33% in men and 50% in women, increasing considerably with age, with cervical pain being one of the main conditions, estimating that 80% of the population has experienced cervicalgia at some time. lifetime. The main symptom is neck pain and restriction of movement, mainly affecting the mobility of the upper cervical region. Although there are studies evaluating the effectiveness of manual techniques, there are currently no studies evaluating the effects on cervical muscle activity and pressure threshold. Therefore, the objective of the present investigation is to evaluate the immediate effects of a manual therapy technique on the threshold pressure of muscular trigger points and on the muscular activity of the upper cervical region in patients with chronic pain and restriction of cervical mobility. higher.

Methods: Clinical trial, randomized, prospective, double-blind study (patient and evaluator). The participants (21 subjects) were divided into 2 groups. The control group will receive a C0-C0 placebo mobilization technique and the experimental group will receive the C0-C1 mobilization technique. In both groups the technique will be carried out by mobilization cycles of 15 seconds and 3 seconds of rest for a total period of 5 min. Pressure threshold, activation of the superficial deep musculature and articular range of the upper cervical region will be measured.

DETAILED DESCRIPTION:
Most cases of pain in the neck region are of mechanical origin. In Spain, its annual prevalence has been estimated to range between 16.7% and 75.1% 2. In Chile, the prevalence is estimated to be 30% in Men and 50% in women, increasing as age increases. It is estimated that, of these cases, 44% have a duration of 6 months or more, giving rise to difficulties not only at work but also in daily life, at home, economically, even in emotional aspects.

The most common symptom is pain in the neck region, which may be associated with restricted movement, dizziness, and manifestations of stress. A large proportion of movement of the cervical spine takes place in the C1-C2 segment, where up to 50% of the total rotation of the cervical spine occurs. There are several techniques to restore cervical mobility, but few of them comply with the guidelines of the IFOMPT (International Federation of Manual Orthopedic Therapists) on the safety and efficacy in the treatment of hypomobility of the upper cervical spine, avoiding positions at the end of the cervical range of motion, especially rotation and extension, and there is also limited scientific evidence of its effectiveness.

The C0-C1 dorsal mobilization technique complies with these recommendations and have been used in previous studies, although there is no evidence of its effects on range of motion, activation of deep cervical musculature and pressure threshold in patients with chronic mechanical cervicalgia. Therefore, the objective of the present investigation is to determine the effects of the dorsal mobilization technique of the atlanto-occipital joint (C0-C1) as adjuvant treatments for Kinesitherapy in users with chronic cervical pain of mechanical origin and rotation deficit in the upper cervical spine.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and over
* Chronic cervical pain
* Sign the informed consent form

Exclusion Criteria:

* History of cervical trauma (Sprains, fracture and / or dislocation of cervical joints)
* Subjects with administration of pain relievers, opiates or muscle relaxants
* Inability to tolerate the supine position
* Subjects with vertiginous syndrome
* Subjects with cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2020-04-10 (Actual); Primary Completion 2020-05-20 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Changes in grade of range of motion of the cervical spine in patients with chronic neck pain | pre-intervention/immediately after the intervention
  The procedure consists of evaluating the cervical flexion, extension, inclination and rotation ranges. The final record will correspond to the average of two measurements on one side and on the contralateral side. The range of motion will be measured with a goniometer

SECONDARY OUTCOMES:
Changes in muscle pressure threshold, measured in kilograms, in patients with chronic neck pain | pre-intervention/immediately after the intervention
  Minimum subject pressure perceived as painful when applied gradually and increasing. This variable is evaluated using an algometer measured in kilograms of pressure.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad San Sebastián, Concepción, Chile